CLINICAL TRIAL: NCT06499636
Title: In Vitro Models Derived From Pediatric Glial Tumors and Pediatric Embryonal Tumors for Drug Testing and Molecular Studies
Brief Title: In Vitro Models From Pediatric Brain Tumors
Acronym: PBTS23
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6351
Record Dates: First submitted 2024-07-08; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Glioma, Malignant; Ependymoma; Medulloblastoma
MeSH Terms: conditions — Glioma; Ependymoma; Medulloblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: other — other

SUMMARY:
Tumors of the Central Nervous System (CNS) represent the leading cause of cancer-related deaths in children. Current treatment options are not curative for most malignant histologies, and intense preclinical and clinical research are necessary to develop more effective therapeutic interventions against these tumors, most of which meet the FDA definition for orphan diseases. The majority of malignant CNS tumors in children and adolescents belong to two broad histologic tumor entities: those of glial origin, such as high-grade glioma (HGG)and ependymoma (EPN), and those of neuronal origin, also identified as embryonal tumors, that include medulloblastoma and AT/RT(1). Over the last few years, whole-genome sequencing, gene-expression profiling and genome-wide methylation studies have greatly deepened our understanding of the biology and genetics of these tumors, allowing for robust stratification in clinically relevant molecular subgroups. The advancement of single-cell omics over the last decade have highlighted the enormous heterogeneity of tumors, a complex mixture of co-existing cancer subclones and supportive normal cell populations.

However, current treatments have remained largely static, and 5-year survival rate for children with malignant CNS tumors only achieves a modest 57.5%.

More effective treatment strategies should include novel chemotherapeutic agents that take into account high intrinsic tumor heterogeneity as well as the complex regulations of transcriptional and translational mechanisms that control protein expression. Identification of novel drugs and treatment strategies is further limited by the paucity of appropriate preclinical models, which mirror the molecular characteristics of distinct tumor subgroups.

We propose to establish patient-derived in vitro models to predict chemotherapeutic drug sensitivity/resistance in malignant pediatric CNS tumors. Next, we propose to perform molecular analyses in tissues of pediatric CNS tumors to determine whether in vitro findings have clinical correlates.

ELIGIBILITY:
Inclusion Criteria:

* Children and young adults who undergo standard surgical resection for suspected primary brain tumors or recurrent brain tumors
* signed written informed consent

Exclusion Criteria:

* no informed consent

Ages: 1 Year to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and young adults
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
1) Establishment of in vitro models derived from pediatric tumors of the CNS, which more faithfully mirror the molecular features and heterogeneity of pediatric EPNs. | 48 months
  Collection and storage of snap-frozen pediatric brain tumor samples (tumor specimens and blood samples).
  Generation of patient-derived cell lines.

SECONDARY OUTCOMES:
2) Preclinical drug testing, to explore the chemotherapeutic potential of selected standard and molecularly-targeted agents. | 24 months
  The models that will be prospectively established in the objective number 1 and the already commercially available models will be used for preclinical in vitro studies with agents belonging to imipridones and DHODH inhibitors
3) Molecular studies on pediatric brain tumor tissues, to determine whether the cellular, molecular and biochemical findings in in vitro models have clinical correlates. | 36 months
  To determine whether the findings in preclinical models have clinical correlates, tumor samples that will prospectively be collected and stored in the Biobank of Fondazione Policlinico Universitario Gemelli will be analyzed for the expression of selected biomarkers. RNA extraction, reverse transcription and real-time PCR will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ruggiero, prof, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Pediatric Oncology Unit- Fondazione Policlinico Gemelli IRCCS, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No